CLINICAL TRIAL: NCT03690427
Title: Investigating the Cardiovascular Toxicity of Exposure to Electronic Hookah Smoking
Brief Title: The Cardiovascular Effects of Electronic Hookah Vaping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mary Rezk-Hanna, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1R21HL145002-01 (NIH); 1R21HL145002-01 (NIH)
Record Dates: First submitted 2018-09-26; First posted 2018-10-01 (Actual); Results first posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-07

CONDITIONS: Endothelial Dysfunction; Inflammation; Oxidative Stress
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: Charcoal-heated hookah smoking vs. electronic hookah vaping
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Charcoal-Heated Hookah followed by Electronic Hookah (Experimental): Participants were invited to smoke a 30-minute traditional charcoal-heated hookah-smoking session, followed by a 30-minute electronic hookah vaping session.
  To mitigate the impact of carryover effects, the two sessions were separated by a minimum of 7-days.
  Interventions: Other: Traditional hookah smoking; Other: Electronic hookah vaping
- Electronic followed by Traditional Charcoal-Heated Hookah (Experimental): Participants were invited to vape a 30-minute electronic hookah session, followed by a 30-minute traditional charcoal-heated hookah smoking session.
  To mitigate the impact of carryover effects, the two sessions were separated by a minimum of 7-days.
  Interventions: Other: Traditional hookah smoking; Other: Electronic hookah vaping

INTERVENTIONS:
Other: Traditional hookah smoking — Charcoal-heated hookah smoking
  Other Names: Combustible hookah smoking
Other: Electronic hookah vaping — Electronic hookah bowl inhalation

SUMMARY:
Hookah (water-pipe) tobacco smoking has quickly grown to become a major global tobacco epidemic among youth; with electronic (e-) hookahs more recently increasing in popularity especially among young female adults, who endorse marketing claims that these products are a safer alternative to traditional hookah, but scientific evidence is lacking. The study aims to elucidate the comparative effects of traditional hookah smoking vs. e-hookah vaping on human vascular and endothelial function; and examine the role of inflammation and oxidative stress, as likely mechanisms in hookah-related cardiovascular disease pathogenesis.

DETAILED DESCRIPTION:
Hookah (water-pipe) tobacco smoking is rapidly increasing in popularity worldwide. Contributing to this popularity is the unsubstantiated belief that traditional charcoal-heated hookah smoke is detoxified as it passes through the water-filled basin. More recently, electronic (e-) hookahs-containing flavored e-liquid that is heated electrically but inhaled through traditional water-pipes-are increasing in popularity in the United States among young female adults, who endorse marketing claims that these products are even safer than traditional charcoal-heated hookah products. The objective of this project is to investigate the comparative effects of traditional charcoal-heated hookah smoking versus e-hookah vaping on endothelial and vascular function and their mechanistic role in the development of cardiovascular disease. The investigators will test the hypothesis that: 1) in the absence of burning charcoal briquettes and virtually any carbon monoxide (CO) exposure, e-hookah vaping acutely impairs endothelial function and evokes acute central arterial stiffness, opposite from the endothelial function augmentation observed after traditional charcoal-heated hookah smoking, which is likely mediated by the large CO boost emitted from burning charcoal briquettes used to heat the flavored hookah tobacco; and 2) the processes of oxidative stress and inflammation play a pivotal mechanistic role underlying these vascular changes. Accordingly, in a cross-over study comparing traditional hookah smoking to e-hookah vaping, the investigators will assess endothelial function measured by brachial artery flow-mediated dilation and aortic stiffness by pulse wave velocity and augmentation index in 18 young healthy hookah smokers 21-39 years old, before and after ad lib 30-minute smoking/ vaping exposure sessions. To test for oxidative stress mediation, the investigators will determine if any acute impairment in endothelial function after e-hookah can be prevented by intravenous Vitamin C infusion, a potent anti-oxidant. Inflammatory and oxidant biomarkers, as well as smoking exposure biomarkers will be collected before and after the exposure sessions. The results of this proposal: (a) stand to fill in gaps in our mechanistic understanding of the comparative effect of traditional vs. e-hookah bowl on vascular and endothelial function; and (b) help inform policy decisions by the FDA about regulation of hookah products.

ELIGIBILITY:
Inclusion Criteria:

* 21-39 years old hookah smokers: smoked hookah >12x in last 12 months
* no history of illicit drugs or marijuana
* no evidence of cardiopulmonary disease by history/ physical
* no diabetes: fasting blood glucose <100 mg/dl
* BP<140/90mmHg
* resting HR<100 bpm
* BMI<30kg•m2
* no prescription medication

Exclusion Criteria:

* exhaled CO>10 ppm (smoking non-abstinence)
* positive pregnancy test
* psychiatric illness

Ages: 21 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rezk-Hanna M, Gupta R, Nettle CO, Dobrin D, Cheng CW, Means A, Brecht ML, Tashkin DP, Araujo JA. Differential Effects of Electronic Hookah Vaping and Traditional Combustible Hookah Smoking on Oxidation, Inflammation, and Arterial Stiffness. Chest. 2022 Jan;161(1):208-218. doi: 10.1016/j.chest.2021.07.027. Epub 2021 Jul 21. PMID 34298007
- [Derived] Rezk-Hanna M, Seals DR, Rossman MJ, Gupta R, Nettle CO, Means A, Dobrin D, Cheng CW, Brecht ML, Mosenifar Z, Araujo JA, Benowitz NL. Ascorbic Acid Prevents Vascular Endothelial Dysfunction Induced by Electronic Hookah (Waterpipe) Vaping. J Am Heart Assoc. 2021 Feb;10(5):e019271. doi: 10.1161/JAHA.120.019271. Epub 2021 Feb 20. PMID 33615833

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through advertisements posted at Southern California colleges and universities, as well as social media websites, from December 2018 to August 2020.
Groups:
- Traditional Followed by Electronic Hookah: Participants were invited to smoke a 30-minute traditional charcoal-heated hookah-smoking session, followed by a 30-minute electronic hookah vaping session.
  To mitigate the impact of carryover effects, the two sessions were separated by a minimum of 7-days.
- Electronic Followed by Traditional Hookah: Participants were invited to vape a 30-minute electronic hookah session, followed by a 30-minute traditional charcoal-heated hookah smoking session.
  To mitigate the impact of carryover effects, the two sessions were separated by a minimum of 7-days.
Period: Overall Study
Arm/Group | Traditional Followed by Electronic Hookah | Electronic Followed by Traditional Hookah
Started | 9 | 10
Completed | 9 | 8
Not Completed | 0 | 2
Not completed — Requested by subject not to complete traditional hookah | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to either smoke hookah first followed by vape hookah or vape hookah first followed by smoke hookah.
Arm/Group | All Study Participants
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Flow-Mediated Dilation (FMD)
Description: Using ultrasound, FMD of the brachial artery induced by reactive hyperemia, was used to measure endothelium-dependent vasodilator function. Baseline diameter and velocity were recorded for 45 seconds and resumed 30 seconds before cuff deflation and continuously for 2 minutes after deflation to obtain true peak vasodilatory response.
Time Frame: Pre- and post- the 30-minute smoking or vaping exposure sessions
Population: All study participants who completed study visits (1 participant had suboptimal ultrasound images from the e-hookah group; and 2 did not have images from the traditional hookah group)
Measure: Mean (Standard Error); unit: percentage of arterial diameter
Groups:
- Electronic Hookah: Participants who completed a 30-minute e-hookah vaping session
- Traditional Hookah: Participants who completed a 30-minute combustible hookah smoking session
Arm/Group | Electronic Hookah | Traditional Hookah
Number analyzed (Participants) | 18 | 17
percentage of arterial diameter
  FMD before exposure session | 6.11 (0.66) | 5.89 (1.02)
  FMD after exposure session | 4.79 (0.58) | 7.31 (0.82)

2. Primary Outcome: Carotid-Femoral Pulse Wave Velocity (Cf-PWV)
Description: Using applanation tonometry, cf-PWV was used to measure central arterial stiffness.
Time Frame: Pre- and post- the 30-minute smoking or vaping exposure sessions
Population: All study participants who completed study visits (unable to obtain data on 4 participants in the e-hookah group)
Measure: Mean (Standard Error); unit: m/sec
Arm/Group | Electronic Hookah | Traditional Hookah
Number analyzed (Participants) | 13 | 17
m/sec
  cf-PWV before exposure session | 8.20 (0.26) | 8.15 (0.20)
  cf-PWV after exposure session | 8.94 (0.33) | 8.71 (0.23)

3. Primary Outcome: HDL Oxidant Index (HOI)
Description: Capacity was determined as the ability of HDL to inhibit LDL-induced oxidation of dihydrodichlorofluorescein into the fluorescent dichlorofluorescein. Capacity was expressed as an HDL oxidative index, determined by the ratio of dichlorofluorescein fluorescence in the presence and absence of HDL. An index of < 1.0 denotes protective antioxidant HDL, whereas an index of > 1.0 indicates pro-oxidant HDL.
Time Frame: Pre- and post- the 30-minute smoking or vaping exposure sessions
Population: All study participants who completed study visits (unable to obtain data on 4 participants in the e-hookah group)
Measure: Mean (Standard Error); unit: index
Arm/Group | Electronic Hookah | Traditional Hookah
Number analyzed (Participants) | 13 | 17
index
  HOI before exposure session | 0.57 (0.05) | 0.56 (0.06)
  HOI after exposure session | 0.58 (0.06) | 0.52 (0.05)

4. Primary Outcome: Paraoxonase-1 (PON-1) Activity
Description: PON-1 activity was determined by the ability of PON-1, associated with HDL, to hydrolyze paraoxon substrate. The hydrolysis of paraoxon (diethyl-p-nitrophenyl phosphate) to p-nitrophenol by PON-1 was determined by incubating 5 mL of plasma with 1.0 mM paraoxon in 100 mM tris-HCl buffer (pH, 8.5).
  Unit of Measure: expressed as micromoles of p-nitrophenol formed per minute for every 1 mL plasma.
Time Frame: Pre- and post- the 30-minute smoking or vaping exposure sessions
Population: All study participants who completed study visits (unable to obtain data on 4 participants in the e-hookah group)
Measure: Mean (Standard Error); unit: units/mL:see Outcome Measure Description
Arm/Group | Electronic Hookah | Traditional Hookah
Number analyzed (Participants) | 13 | 17
units/mL:see Outcome Measure Description
  PON-1 before exposure session | 1071.24 (188.79) | 709.32 (112.43)
  PON-1 after exposure session | 1151.73 (207.98) | 701.29 (110.67)

5. Primary Outcome: Arylesterase Activity
Description: Arylesterase activity (lipid peroxidation biomarker) was determined by the rate of hydrolysis of phenyl acetate to phenol. Briefly, 4 mL plasma was incubated with 3.5 mM phenyl acetate in 9 mM Tris-HCl buffer (pH, 8.0) containing 0.9 mM CaCl2 at RT. The kinetics of phenol formation were determined by recording the absorbance at 270 nm every 15 s for 2 min.
  Unit of Measure: nanomoles of product formed per minute per milliliter of plasma.
Time Frame: Pre- and post- the 30-minute smoking or vaping exposure sessions.
Population: All study participants who completed study visits (unable to obtain data on 1 participant from the e-hookah group and 3 participants from the traditional hookah group).
Measure: Mean (Standard Error); unit: units/mL:see Outcome Measure Description
Arm/Group | Electronic Hookah | Traditional Hookah
Number analyzed (Participants) | 16 | 14
units/mL:see Outcome Measure Description
  Arylesterase activity before exposure session | 277.36 (14.26) | 281.38 (19.33)
  Arylesterase activity after exposure session | 295.78 (16.78) | 285.06 (16.78)

6. Primary Outcome: High-sensitivity C-reactive Protein (Hs-CRP) Levels
Description: Plasma hs-CRP (inflammatory biomarker)
Time Frame: Pre- and post- the 30-minute smoking or vaping exposure sessions
Population: All study participants who completed study visits (unable to obtain data on 2 participants in the traditional hookah group)
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Electronic Hookah | Traditional Hookah
Number analyzed (Participants) | 17 | 15
mg/L
  hs-CRP before exposure session | 0.72 (0.12) | 0.77 (0.19)
  hs-CRP after exposure session | 0.76 (0.13) | 0.77 (0.19)

7. Primary Outcome: Tumor Necrosis Factor-α (TNFα) Concentrations
Description: Plasma TNFα (inflammatory biomarker)
Time Frame: Pre- and post- the 30-minute smoking or vaping exposure sessions
Population: All study participants who completed study visits (unable to obtain data on 1 participant in the e-hookah group)
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Electronic Hookah | Traditional Hookah
Number analyzed (Participants) | 16 | 17
pg/mL
  TNFα before exposure session | 0.69 (0.06) | 0.85 (0.08)
  TNFα after exposure session | 0.76 (0.08) | 0.82 (0.08)

8. Secondary Outcome: Flow-Mediated Dilation (FMD)
Description: Using ultrasound, FMD of the brachial artery, induced by reactive hyperemia, was used to measure endothelium-dependent vasodilator function after intravenous infusion of antioxidant ascorbic acid. Infusion of antioxidant ascorbic acid was done before the e-hookah vaping session.
Time Frame: Effect of FMD with e-hookah vaping examined after pretreatment of intravenous infusion of antioxidant ascorbic acid (administered over 60 minutes at 0.5 mL min-1)
Population: A subset of participants, who completed the e-hookah vaping protocol.
Measure: Mean (Standard Error); unit: percentage of arterial diameter
Groups:
- Electronic Hookah: Assess the acute effects of e-hookah vaping on FMD before and after intravenous administration of a supra-physiological dose of ascorbic acid.
Arm/Group | Electronic Hookah
Number analyzed (Participants) | 11
percentage of arterial diameter
  FMD before e-hookah vaping | 9.46 (0.87)
  FMD after e-hookah vaping | 8.74 (0.84)

9. Secondary Outcome: Endothelium-independent Vasodilator Function (Control Test for Endothelium-dependent Vasodilator Function)
Description: As a control test for the assessment of endothelium-dependent vasodilator function, using ultrasound the brachial artery, endothelium-independent dilatation was assessed by administering sublingual nitroglycerin. This measure was assessed 10 minutes after FMD testing. Ultrasound images were recorded continuously for a total of 10 minutes
Time Frame: Pre- and post- sublingual administration of nitroglycerin (0.15 mg), which was administrated before and after e-hookah vaping.
Population: A subset of participants, who completed the e-hookah vaping protocol.
Measure: Mean (Standard Error); unit: percentage of arterial diameter
Arm/Group | Electronic Hookah
Number analyzed (Participants) | 8
percentage of arterial diameter
  Dilation before e-hookah vaping | 27.15 (1.98)
  Dilation after e-hookah vaping | 25.17 (1.87)

10. Secondary Outcome: Augmentation Index (AI)
Description: AI was used to measure central stiffness. It was calculated as the ratio of augmentation pressure (difference between the second and first systolic peaks of the aortic pressure waveform) and pulse pressure expressed as a percentage.
Time Frame: Pre- and post- the 30-minute smoking or vaping exposure sessions
Population: All study participants who completed study visits (unable to obtain data on 4 participants in the e-hookah group and 1 in the traditional hookah group)
Measure: Mean (Standard Deviation); unit: percentage of the pulse pressure
Arm/Group | Electronic Hookah | Traditional Hookah
Number analyzed (Participants) | 13 | 16
percentage of the pulse pressure
  AI before exposure session | 7.97 (2.97) | 7.79 (2.54)
  AI after exposure session | 13.55 (3.24) | 10.66 (2.98)

11. Secondary Outcome: Interleukin 6 (IL-6) Levels
Description: Plasma IL-6 (inflammatory biomarker).
Time Frame: A change between two points is reported below (e.g., value at post-exposure session minus value at pre-exposure session).
Population: All study participants who completed study visits (unable to obtain data on 5 participants in the e-hookah group)
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Electronic Hookah | Traditional Hookah
Number analyzed (Participants) | 12 | 17
pg/mL | 0.13 (0.08) | 0.04 (0.06)

12. Secondary Outcome: Interleukin 10 (IL-10) Levels
Description: Serum IL-10 (anti-inflammatory biomarker)
Time Frame: as for outcome 11
Population: All study participants who completed study visits (unable to obtain data on 5 participants in the e-hookah group)
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Electronic Hookah | Traditional Hookah
Number analyzed (Participants) | 12 | 17
pg/mL | 0.03 (0.03) | -0.01 (0.01)

13. Secondary Outcome: Nicotine Levels
Description: Plasma nicotine levels (smoking or vaping exposure biomarker)
Time Frame: Pre- and post- the 30-minute smoking or vaping exposure sessions
Population: All study participants who completed study visits (unable to obtain data on 1 participant in the e-hookah group and 1 participant in the traditional hookah group)
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Electronic Hookah | Traditional Hookah
Number analyzed (Participants) | 16 | 16
ng/mL
  Plasma nicotine before exposure session | 0.59 (0.09) | 0.82 (0.24)
  Plasma nicotine after exposure session | 5.83 (0.96) | 6.96 (1.11)

14. Secondary Outcome: Carbon Monoxide (CO) Levels
Description: Exhaled CO levels (smoking or vaping exposure biomarker)
Time Frame: Pre- and post- the 30-minute smoking or vaping exposure sessions
Population: All study participants who completed study visits (unable to obtain data on 1 participant in the e-hookah group; and 1 participant in the traditional hookah group)
Measure: Mean (Standard Error); unit: ppm
Arm/Group | Electronic Hookah | Traditional Hookah
Number analyzed (Participants) | 16 | 16
ppm
  CO before exposure session | 2.58 (0.27) | 3.38 (0.49)
  CO after exposure session | 2.31 (0.20) | 40.19 (6.69)

ADVERSE EVENTS:
Time Frame: Throughout the entire study duration (i.e., scheduled study visit lasting 4-5 hours), including the 30-minute hookah smoking and e-hookah vaping exposure sessions.
Groups:
- Traditional Hookah: Participants who were invited to smoke a 30-minute combustible charcoal-heated hookah-smoking session.
- Electronic Hookah: Participants who were invited to vape a 30-minute electronic hookah bowl session.
Arm/Group | Traditional Hookah | Electronic Hookah
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/19
Other Adverse Events (participants affected / at risk) | 0/17 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT03690427/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT03690427/SAP_001.pdf